CLINICAL TRIAL: NCT02008253
Title: Intrastromal Corneal Ring Segment Implantation for Ectasia After Refractive Surgery
Brief Title: Intrastromal Corneal Ring for Ectasia After Refractive Surgery (Anel)
Status: Completed | Type: Observational
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Sponsor
Other Study IDs: BQ-1-14 - ARVO
Record Dates: First submitted 2013-12-01; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Ectasia
Keywords: INTRASTROMAL CORNEAL RING; ASTIGMATISM
MeSH Terms: conditions — Dilatation, Pathologic; Astigmatism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- INTRASTROMAL CORNEAL RING SEGMENT: Forty-two eyes of 26 patients, 14 men and 12 women, with ectasia after refractive surgery were studied in a nonrandomized, retrospective, observational case series.
  Interventions: Procedure: INTRASTROMAL CORNEAL RING SEGMENT

INTERVENTIONS:
Procedure: INTRASTROMAL CORNEAL RING SEGMENT — Corneal tunnels were created by means of mechanical dissection in all eyes. Main outcome measures included UCVA, BCVA, refraction, keratometry and computerized analysis of corneal topography.

SUMMARY:
To evaluate the clinical outcomes of intrastromal corneal ring segment (ICRS) implantation to correct keratoconus on eyes with prior refractive surgery.

DETAILED DESCRIPTION:
Forty-two eyes of 26 patients, 14 men and 12 women, with ectasia after refractive surgery were studied in a nonrandomized, retrospective, observational case series. Mean age at the time of ICRS implantation was 30,5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients 19 to 48 years old
* Keratoconus (ectasia) on eyes with prior refractive surgery

Exclusion Criteria:

* Diabetes
* Autoimmune diseases

Ages: 19 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients residents in Brazil with ectasia after refractive surgery
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2010-04; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Intrastromal Corneal Ring Segment Implantation for Ectasia After Refractive Surgery | Mean follow-up after ICRS implantation was 12 months (range, 09 to 22 months).
  To evaluate the clinical outcomes of intrastromal corneal ring segment (ICRS) implantation to correct keratoconus on eyes with prior refractive surgery. Corneal tunnels were created by means of mechanical dissection in all eyes. Main outcome measures included UCVA, BCVA, refraction, keratometry and computerized analysis of corneal topography.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Rossana S Stival, Study Chair — Instituto de Olhos de Goiânia
Locations (1):
- Instituto de Olhos de Goiânia, Goiânia, Goiás, Brazil